CLINICAL TRIAL: NCT02920710
Title: ACTHAR Therapy for Central Nervous System Sarcoidosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: The Cleveland Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTHAR CNS
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: H.P. Achtar Gel 80 U (Experimental): H.P. Acthar Gel (repository corticotropin) Injection, 80 U daily for 10 days, then 80 U twice weekly for up to a total of 48 weeks on therapy.
  Interventions: Drug: Repository Corticotropin Injection

INTERVENTIONS:
Drug: Repository Corticotropin Injection — * Initial treatment with 80 units daily for ten days (induction phase)
  * Maintenance treatment with 80 units twice weekly (maintenance phase)
  Other Names: H.P. Acthar Gel; ACTH Gel; ACTH

SUMMARY:
There is a need for a more reliable, expeditious therapy that can be used as an alternative to glucocorticoids in severe Central Nervous System (CNS) sarcoidosis. This study aims to provide evidence for effectiveness of ACTHAR gel in CNS sarcoidosis, and provide information about its safety and tolerability

DETAILED DESCRIPTION:
Central nervous system (CNS) involvement is one of the most severe manifestations of sarcoidosis. Sarcoidosis affecting the leptomeninges, spinal cord, or brain parenchyma portends a difficult course and frequently results in severe disability or death (1). Treatment of moderate and severe CNS sarcoidosis typically involves a combination of corticosteroids and cytotoxic agents such as methotrexate (2). Unfortunately, most response rates are reportedly only in the 29-38% range for corticosteroids alone, and the effects of cytotoxic agents in sarcoidosis require up to 6 months to occur. A typical scenario is that patients are treated for prolonged periods with high dose glucocorticoids with suboptimal effectiveness despite development of substantial toxicities. Some series report that cyclophosphamide or infliximab may be beneficial (3), but these approaches are limited by potentially severe toxicities, loss of effectiveness, or payor constraints.

. ACTHAR is a 39-amino acid peptide natural form of adrenocorticotropin hormone (ACTH) that was initially approved in 1952 by the FDA. It has since been approved for 19 indications including respiratory sarcoidosis, multiple sclerosis, and infantile spasms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sarcoidosis as defined by ATS/ERS/WASOG (American Thoracic Society/European Thoracic Society/World Association for Sarcoidosis and Other Granulomatous Disorders)
* Stable baseline immunosuppressive medications
* Moderate to severe disease as defined by at least one of the following criteria:

  * Cranial nerve palsy
  * Neurologic deficits related to intraparenchymal brain, spinal cord and/or cauda equina involvement
  * Dural or leptomeningeal involvement of brain and/or spinal cord
  * Hydrocephalus
  * Seizures

Exclusion Criteria:

* Diagnosis of any underlying neurologic disorder that would potentially confound interpretation of the study results
* Significant change in corticosteroid dose within the past 4 weeks, or other immunosuppressive medication within the past 6 months
* Evidence of current serious infection, or a history of chronic or recurring infections.
* Contraindication to high-dose corticosteroids (e.g. uncontrolled blood sugar).
* Allergies to pig-derived proteins
* Have a history of any opportunistic infection within 6 months prior to screening
* History of malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinically significant improvement - successful glucocorticoid tapering. | 12 Weeks

SECONDARY OUTCOMES:
Proportion of patients with clinically significant improvement - no need for escalation of other therapy. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Culver, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided